CLINICAL TRIAL: NCT04566900
Title: Enhancing Gamma Band Response in Mild Cognitive Impairment to Improve Working Memory
Brief Title: Neurofeedback to Improve Working Memory in Mild Cognitive Impairment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Fiza Singh, Associate Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192022
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment
Keywords: neurofeedback
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: MCI subjects will be assigned to active intervention or placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-blind, randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Subjects will be given a choice of videos consisting of still images set to music. Whether the video progresses and music continues to play will depend on the subject's ability to maintain frontal gamma oscillatory activity within a prespecified range. Over successive weeks, the parameters for positive feedback (music and video progression) will become incrementally more difficult.
  Interventions: Behavioral: Neurofeedback
- Placebo (Sham Comparator): Video and music progression will be random and will not depend on brain activity. Any progression will be by random chance alone.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Neurofeedback — Neurofeedback is a technique where brain functions are made accessible to the subject in the form of a metaphor. For instance, frontal brain activity may be shown as an airplane flying. Once the activity is made accessible, the subject can modulate it in a pre-specified direction. The parameters used to achieve successful feedback are made difficult over time and hence the brain is taught or conditioned to improve performance.
  Arms: Active Treatment
Other: Placebo — Subjects in this arm will undergo all of the same testing as active treatment. Music and video progression will not depend on brain activity. Instead feedback will be random.
  Arms: Placebo

SUMMARY:
Mild cognitive impairment (MCI) has been identified as an early phase of Alzheimer's disease (AD), a neurodegenerative disorder expected to affect 13.9 million Americans by 2060. AD causes a progressive cognitive decline, including problems related to learning and memory, that adversely affects life quality. Treatment intervention at the MCI stage of the disease could potentially slow down the rate at which people may convert from MCI to AD. Increasing evidence suggests that abnormal activity in frontal regions of the brain is associated with cognitive deficits observed in AD. Furthermore, previous research has shown that neurofeedback (NFB) training targeting these regions can improve memory, making it a potential treatment for AD. NFB is a technique where an individual learns to change his/her brain function in a particular direction, once that function has been made accessible through a visual or auditory metaphor. We are proposing a novel, computer-based brain-training program to enhance frontal gamma oscillatory activity in individuals with MCI. Results from this study will build the scientific foundation necessary for larger clinical trials dedicated to improving treatment options and outcomes for patients with MCI.

DETAILED DESCRIPTION:
This is a randomized, double-blind, clinical trial to test the efficacy of gamma-neurofeedback (G-NFB) compared to a placebo (P-NFB) in individuals with MCI. 112 consented participants will be randomized to receive G-NFB (n=56) or placebo-NFB (n=56) during 30-45 minute sessions twice per week for 12 weeks (24 total sessions). Memory and other cognitive domains will be measured using paper and pencil and computerized tests every 4 weeks during the study and at 4 weeks post completion of study.

ELIGIBILITY:
Inclusion Criteria:

1. Meet criteria for mild cognitive impairment (MCI).
2. Living independently.
3. Literate in English.
4. Competent to participate in the informed consent process and provide voluntary informed consent.

Exclusion Criteria:

1. Frontal temporal dementia
2. Active alcohol or substance use disorder within the past year.
3. Brain cancer
4. Stroke within the last 2 years
5. Anti-epileptic medication
6. Prior head injury involving loss of consciousness
7. Seizure disorder
8. Use of medications likely to affect cognitive function (cf. donepezil, memantine). We will not exclude for other medications but will examine their effects and include medications as covariates as appropriate (e.g., presence v. absence; anticholinergic load).
9. The potential benefits of the study do not outweigh the potential risks of the study, as determined by the PI.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Working Memory accuracy | From baseline to 12 weeks of treatment
  Change in the computerized test, N-back will be used to measure working memory.

SECONDARY OUTCOMES:
Durability of Change in Working Memory accuracy | From baseline to 4weeks post end of study
  Change in the computerized test, N-back will be used to measure working memory.
Change in Gamma Band Response | From baseline to 12 weeks of treatment
  Change in Gamma oscillations will be measured while the subject performs the n-back task.
Durability of Gamma Band Response | From baseline to 4weeks post end of study
  Change in Gamma oscillations will be measured while the subject performs the n-back task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California at San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Dohnel K, Sommer M, Ibach B, Rothmayr C, Meinhardt J, Hajak G. Neural correlates of emotional working memory in patients with mild cognitive impairment. Neuropsychologia. 2008 Jan 15;46(1):37-48. doi: 10.1016/j.neuropsychologia.2007.08.012. Epub 2007 Aug 23. PMID 17915264
- [Background] Leuchter AF, Newton TF, Cook IA, Walter DO, Rosenberg-Thompson S, Lachenbruch PA. Changes in brain functional connectivity in Alzheimer-type and multi-infarct dementia. Brain. 1992 Oct;115 ( Pt 5):1543-61. doi: 10.1093/brain/115.5.1543. PMID 1422803
- [Background] Uhlhaas PJ, Singer W. Neural synchrony in brain disorders: relevance for cognitive dysfunctions and pathophysiology. Neuron. 2006 Oct 5;52(1):155-68. doi: 10.1016/j.neuron.2006.09.020. PMID 17015233
- [Background] Stam CJ, van Cappellen van Walsum AM, Pijnenburg YA, Berendse HW, de Munck JC, Scheltens P, van Dijk BW. Generalized synchronization of MEG recordings in Alzheimer's Disease: evidence for involvement of the gamma band. J Clin Neurophysiol. 2002 Dec;19(6):562-74. doi: 10.1097/00004691-200212000-00010. PMID 12488788

DOCUMENTS (1):
  • Informed Consent Form (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT04566900/ICF_001.pdf